CLINICAL TRIAL: NCT01789294
Title: CLINICAL MANAGEMENT OF CHILDHOOD INTESTINAL LYMPHOID NODULAR HYPERPLASIA: A RANDOMIZED CONTROLLED CLINICAL TRIAL.
Brief Title: Clinical Management of Childhood Intestinal Lymphoid Nodular Hyperplasia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ped-LNH
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2008-11

CONDITIONS: Intestinal LNH
Keywords: lymphoid nodular hyperplasia; food allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Mesalamine; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mesalamine (Experimental): A standard 50 mg/kg/die daily dose of oral mesalamine was prescribed by Pediatric Gastroenterologists, which informed parents of potential side effects
  Interventions: Drug: Mesalamine
- Observation (No Intervention): A close clinical observation without therapy was taken in control patients, whom parents were alerted to refer immediately if symptoms persisted or get worse.
- DIET (Experimental): Dietetic avoidance of cow's milk and egg, plus foods eventually detected by skin tests, was prescribed by Pediatric Allergologists
  Interventions: Behavioral: DIET

INTERVENTIONS:
Drug: Mesalamine — A standard 50 mg/kg/die daily dose of oral mesalamine was prescribed by Pediatric Gastroenterologists, which informed parents of potential side effects. Whether the drug was not well tolerated, patients were drop out. Treatment was discontinued at time 1 to look for symptom recurrence.
  Arms: Mesalamine
Behavioral: DIET — Dietetic avoidance of cow's milk and egg, plus foods eventually detected by skin tests, was prescribed by Pediatric Allergologists. To ensure the correct adherence to diet with no nutritional impairment, a scheme of admitted foods and an appropriate calcium supplement dose were given to patients.
  Arms: DIET

SUMMARY:
Aim of this prospective, parallel multi-arm, randomized, clinical trial, was to compare the clinical outcome of patients Methods.We recruited children who undergone diagnostic colonoscopy in Umberto I Pediatric Department (Rome, Italy) from 2008 to 2010. Eligibility criteria were: 1) only demonstration of LNH; 2) no concomitant disease; 3) no treatment assumed since the clinical onset. Patients were allocated 1:1:1 to dietetic (Group A) vs mesalamine (Group B) vs no treatment (Group C) for a 8-weeks period. Skin prick tests and patch test for common foods, and symptoms scoring at baseline and follow up have been performed by blinded clinicians. Chi-square test for trend was used to compare the frequency of symptoms score improvement (>1 point) among groups. The association of baseline features of patients with the clinical response was estimated by frequency analysis.

DETAILED DESCRIPTION:
Lymphoid nodular hyperplasia (LNH) of the lower gastrointestinal tract is a common finding in pediatric colonoscopies, whose clinical significance is not yet been clearly established. Although initially considered to be a normal, age-related variant, some authors recently suggested to regard LNH as a marker of food allergy (FA).

ELIGIBILITY:
Inclusion Criteria:

1. isolated finding of LNH[18], defined as the demonstration of a significant cluster of lymphoid nodules (>10/visible field) by endoscopy and lymphoid follicle hyperplasia by hystology;
2. negative results of preliminary evaluation

Exclusion Criteria:

1. diagnosis of concomitant inflammatory, rheumatic or infectious disease, and
2. the assumption of any dietetic or therapy since the clinical onset.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 8 weeks
  to identify an appropriate management approach for LNH by evaluation of clinical severity and response.
  Clinical severity at time 0 and 1 was assessed by Pediatric Gastroenterologists blinded to allocation concealment. Basing on standardized Childhood behaviour checklists questionaire compiled by parents, symptoms were graded using a validated score of abdominal pain (from 0 to 12).
  Clinical response was defined as the improvement of at least 1 point in symptom scores from time 0 to 1.

SECONDARY OUTCOMES:
predictive factors | 8 weeks
  we evaluated whether symptoms severity, site of LNH, presence of food sensitization and predisposition to atopy, should be predictive for the clinical response

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Pediatrics, Sapienza - University of Rome, Rome, Italy